CLINICAL TRIAL: NCT01345383
Title: Impact of Current Smoking in the Tolerance of Bronchoscopy
Status: Terminated | Type: Observational
Why Stopped: the physician responsable for this protocol left our hospital
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Chef de clinique adjoint, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: AK/10-05-3898/38
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Smokers
Keywords: smoking; bronchoscopy; cough
MeSH Terms: conditions — Smoking; Cough | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Current smokers
  Interventions: Procedure: bronchoscopy

INTERVENTIONS:
Procedure: bronchoscopy — Routine bronchoscopy under local anesthesia (lidocain). Duration: +/- 10 min

SUMMARY:
The purpose of this study is to study the impact of smoking in the preceding hours before a bronchoscopy on the tolerance of this exam.

DETAILED DESCRIPTION:
Tolerance evaluation of the bronchoscopy on current and regular smokers. The investigators assess episodes of cough, dyspnea, volume of lidocain (liquid 1% and in spray 10%), duration of the procedure, episodes of desaturation and completion of the bronchoscopy.

The investigators compare patients who did not smoke in the 6 hours before the bronchoscopy and those who have smoked.

ELIGIBILITY:
Inclusion Criteria:

* current and regular smoker
* bronchoscopy under local anesthesia

Exclusion Criteria:

* patients needing EBUS or fluoroscopy
* intravenous sedative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current and regular smokers needing a bronchoscopy as determined by their own physician
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
cough | Day 1
  number of cough episodes during the bronchoscopy

SECONDARY OUTCOMES:
dyspnea | day 1
  dyspnea evaluation before and during the bronchoscopy
Lidocaine volume | day 1
  Volume of local anesthesic needed during bronchoscopy
length of bronchoscopy | Day 1
  length of bronchoscopy
desaturation episodes | day 1
  desaturation episodes during bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle De Meulder, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHU Saint Pierre, Brussels, Belgium